CLINICAL TRIAL: NCT05788172
Title: Quantifying Menstrual Blood Loss: Validating the Methodology for Stable Iron Isotopes Dilution Against the Alkaline Hematin Method
Brief Title: Measuring Menstrual Iron Loss Using the Iron Isotope Dilution Technique
Acronym: MBL_Loss
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Wageningen University and Research (Other); Sight and Life Foundation (Unknown); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Principal Investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: MBL_Loss
Record Dates: First submitted 2023-01-30; First posted 2023-03-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Iron-deficiency; Menorrhagia; Anemia
Keywords: anemia; menstruation; alkaline hematin; iron isotope dilution; blood loss; menorrhagia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Menorrhagia; Anemia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for the measurement of hemoglobin, iron status and iron isotope dilution, as well as menstrual iron loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Female 18-30 year olds, who have already been labelled with stable iron isotopes at least 12 months prior to study start.
  Interventions: Other: Iron isotope dilution; Other: Alkaline hematin method

INTERVENTIONS:
Other: Iron isotope dilution — Menstrual blood loss will be determined using the iron isotope dilution technique and compared to the amount determined via the alkaline hematin method.
Other: Alkaline hematin method — Menstrual blood loss will be determined using the alkaline hematin method and compared to the amount determined via the iron isotope dilution technique.

SUMMARY:
It is very difficult to quantify menstrual blood loss, the reference method is a tedious one. This is a problem, as it is not conducive to objectively measuring menstrual blood loss and understanding the contribution of menstrual iron loss to iron deficiency anemia. With this study, the investigators aim to investigate iron loss during the menstrual cycle and aim to validate a much simpler technique.

DETAILED DESCRIPTION:
Anemia reduction efforts have largely focused on increasing iron intakes such as improving diet quality, food fortification with iron, iron supplementation, biofortification. There is little information on the contribution of menstrual iron loss to iron deficiency anemia.

Indeed, the accurate measurement of menstrual blood loss volume and iron loss is difficult. Self-perception of heavy menstrual blood loss poorly predicts actual blood loss, and the objective measurement of menstrual blood loss remains a tedious method. Various methods have been used to objectively measure menstrual blood loss volume including radioisotopes, but these methods are invasive. The investigators aim to validate a much simpler technique, namely the stable iron isotope dilution methodology. This is a promising new method for quantifying long-term body iron balance, absorption, and loss which has not been applied previously to measure menstrual iron losses. Validating this new method against the alkaline hematin reference method would be an important step to encourage menstrual blood loss measurements and shed light on the contribution of menstrual blood loss to iron deficiency and iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-30 years old
* Already labelled with stable iron isotopes at least 12 months prior to study start
* Weight <70 kg
* Normal body mass index (18.5 - 25kg/m2)
* Regular menstrual cycle (self-reported cycle length between 28 and 35 days in the past 6 months)
* Signed informed consent
* Able to read and understand English

Exclusion Criteria:

* Use of hormonal contraceptives within a 3-month recall period
* Anemia (hemoglobin < 117 g/L)
* Any known major metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer, or cardiovascular diseases (according to the participants own statement)
* Women with severe menstrual cramps
* Consumption of iron-containing supplements within 1 month prior to the start of study
* Known difficulties with blood sampling
* Pregnancy (serum human chorionic gonadotropin (hCG) < 5 mIU/mL)
* Current smoking (>1 cigarette per week over a 1-month recall period)
* Women who are planning to get pregnant
* Inability to follow the study protocol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female 18-30 year olds, who have already been labelled with stable iron isotopes.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Amount of menstrual blood lost (mL/cycle) | At the beginning of menstrual cycle 1 (cycle length between 28 and 35 days)
  The amount of menstrual blood lost will be determined using the alkaline hematin reference method. All sanitary material is collected during menstruation in each cycle and the amount of blood lost is measured directly in this material. For each cycle the total amount of blood lost during this cycle is determined (there will be one value only during each cycle).
Amount of menstrual blood lost (mL/cycle) | At the beginning of menstrual cycle 2 (cycle length between 28 and 35 days)
  The amount of menstrual blood lost will be determined using the alkaline hematin reference method. All sanitary material is collected during menstruation in each cycle and the amount of blood lost is measured directly in this material. For each cycle the total amount of blood lost during this cycle is determined (there will be one value only during each cycle).
Amount of menstrual blood lost (mL/cycle) | At the beginning of menstrual cycle 3 (cycle length between 28 and 35 days)
  The amount of menstrual blood lost will be determined using the alkaline hematin reference method. All sanitary material is collected during menstruation in each cycle and the amount of blood lost is measured directly in this material. For each cycle the total amount of blood lost during this cycle is determined (there will be one value only during each cycle).
Change in isotopic ratio per cycle | Screening, day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78 and 85
  The change in iron losses between the time of menstruation and the remaining duration of the cycle will be measured based on the dilution of the stable iron isotopes in the blood

SECONDARY OUTCOMES:
Hemoglobin concentration (g/L) | Screening, day 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78 and 85
  Hemoglobin will be measured to determine the presence of anemia and for the standardization of menstrual blood loss measurement
Serum ferritin (microg/L) | Day 1 and 85
  Iron status parameter
Serum transferrin receptor (mg/L) | Day 1 and 85
  Iron status parameter
Alpha-1-acid glycoprotein (g/L) | Day 1 and 85
  Chronic inflammation parameter
C-reactive protein (mg/L) | Day 1 and 85
  Acute inflammation parameter

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, PhD, Principal Investigator — ETH
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No